CLINICAL TRIAL: NCT05025137
Title: Comparing the Effectiveness of Flexi-Bar and Multi-Component Exercises on Improving the Frailty, Physical Fitness, and Musculoskeletal Discomfort of Older Adults: a Randomized Controlled Trial
Brief Title: Flexi-Bar and Multi-Component Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Shang-Yu (Other)
Responsible Party: Sponsor-Investigator, Yang Shang-Yu, Assistant professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRREC-109
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexi-Bar group (Experimental): Participants in the Flexi-Bar group performed a 60-minute Flexi-Bar exercise every week for 12 consecutive weeks.
  Interventions: Other: Flexi-Bar Exercise
- Multi-Component exercise group (Experimental): Participants in the Multi-Component exercise group performed a 60-minute Multi-Component exercise every week for 12 consecutive weeks.
  Interventions: Other: Multi-Component exercise

INTERVENTIONS:
Other: Flexi-Bar Exercise — In the experimental group, the Flexi-Bar was adopted as the tool for active vibration exercises. Featuring light weight and ease of operation, it weighs only 460 grams and has a vibration frequency of 4-5 Hz. With diversified functions, the Flexi-Bar can improve posture, burn fat, strengthen connective tissue, enhance body shape, and increase muscle strength.
  The 12-week Flexi-Bar exercise course in this study was created by two assistant professors specializing in rehabilitation (one with an occupational therapy certificate and the other with a physical therapy certificate). The course, composed of one 60-minute class per week for a total of 12 weeks, progressed gradually from basic activities (e.g., standing with both feet) to advanced activities (e.g., standing with one foot).
  Arms: Flexi-Bar group
Other: Multi-Component exercise — Alternatively, in the control group, the Multi-Component exercise was adopted, which included aerobic, resistance, flexibility, and balance exercises. The course was composed of one 60-minute class per week for a total of 12 weeks. The design was based on the ACSM's recommendations for the multiple-component exercise of the elderly (Chodzko-Zajko et al., 2009) and videos of the National Health Exercises for the Elderly formulated by the Ministry of Health and Welfare (Ministry of Health and Welfare, 2017). The course was created and led by a physical therapist to gradually progress from sitting postures to standing and walking postures. Additionally, the intensity of the exercises was adjusted according to the participants' physical conditions; fitness equipment was introduced when appropriate.
  Arms: Multi-Component exercise group

SUMMARY:
Background: Previous studies have suggested that both Flexi-Bar and Multi-Component exercises can improve an individual's physical fitness and musculoskeletal discomfort. However, determining which is more effective in enhancing the frailty, physical fitness, and musculoskeletal discomfort of the elderly remains controversial.

Objective: This study aims to investigate differences in the effectiveness of Flexi-Bar and Multi-Component exercises in improving the frailty, physical fitness, and musculoskeletal discomfort of the elderly after 12 weeks of intervention.

Methods: A single-blind randomized controlled trial was conducted to collect data from a city in central Taiwan. Participants were randomly divided into a Flexi-Bar group (FB group) and a Multi-Component exercise group (MCE group). Participants in the FB group performed a 60-minute Flexi-Bar exercise every week for 12 consecutive weeks. Meanwhile, Participants in the MCE group performed a 60-minute Multi-Component exercise every week for 12 consecutive weeks. Tests were conducted both before and after the 12-week intervention using items including the Kihon Checklist, Senior Fitness Test, and Nordic Musculoskeletal Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* (1) participants aged 65 years and over;
* (2) participants who could communicate in Mandarin or Taiwanese and cooperate with sports activities; and
* (3) participants who could walk independently without assistance (or with aid).

Exclusion Criteria:

* (1) participants with unstable physiological conditions (or those who were recommended against participating in physical activities by their doctor);
* (2) participants with unstable mental conditions; and
* (3) participants who could not complete the 12-week exercise intervention.

Ages: 65 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Kihon Checklist | 10-15 minutes
  The KCL consists of 25 True or False questions and covers seven aspects, including living independence, exercise function, nutrition, oral function, social interaction, dementia, and depression. The total score of all items, which ranged between 0 and 25, was then used to evaluate the participant's frailty. Participants with a score of 10 and greater were categorized as the frail population. The higher the score, the higher the degree of frailty. The reliability and validity of the Chinese version of the KCL was well verified (Tsay et al., 2018).

SECONDARY OUTCOMES:
Senior Fitness Test | 30-40 minutes
  The SFT was designed by Rikli and Jones (2013) to assess the physical fitness of the elderly in daily activities. It includes six tests, namely (1) chair stand test; (2) arm curl test; (3) 2-minute step test; (4) chair sit-and-reach test; (5) back scratch test; and (6) eight-foot up-and-go test.
Nordic Musculoskeletal Questionnaire | 10-15 minutes
  Developed by Kuorinka et al. (1987), the NMQ asks participants whether they have experienced pain, soreness, numbness, tingling, or any other discomfort in 15 body parts on both sides (including neck, shoulders, upper back, elbows, lower back or waist, hands or wrists, hips or thighs, and knees and ankles or feet). The human body illustration in the questionnaire allows subjects to easily and clearly identify the location of musculoskeletal discomfort. The number of body parts with discomfort is then calculated by adding the number of locations experiencing any discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University, Taichung, WuFeng, Taiwan